CLINICAL TRIAL: NCT06163612
Title: Effect of Suicidality in Major Depressive Disorder During Social Cognition
Brief Title: Effect of Suicidality on Social Cognition
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-333
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Suicide; Major Depressive Disorder
MeSH Terms: conditions — Suicide; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls, or people who do not have depression.
  Interventions: Behavioral: Clinical Interview; Behavioral: Clinical Questionnaires; Other: Brain Scan; Behavioral: Behavioural Games
- People diagnosed with MDD and a history of suicide attempt
  Interventions: Behavioral: Clinical Interview; Behavioral: Clinical Questionnaires; Other: Brain Scan; Behavioral: Behavioural Games
- People diagnosed with MDD without a history of suicide attempt
  Interventions: Behavioral: Clinical Interview; Behavioral: Clinical Questionnaires; Other: Brain Scan; Behavioral: Behavioural Games

INTERVENTIONS:
Behavioral: Clinical Interview — A study team member will meet the participant to ask questions regarding the degree of depression at the beginning of the study. This interview will take approximately 1 hour.
Behavioral: Clinical Questionnaires — A study team member will ask the participant to complete questionnaires assessing the severity of the participant's depression, daily activities, personality/traits, and quality of life. If the participant opts to complete these questionnaires at home, they will be emailed them within 24 hours of this visit. These questionnaires will take approximately 1-2 hours.
Other: Brain Scan — The participant will be asked to undergo a magnetic resonance imaging (MRI) scan to look at the structure and function of their brain. The functional MRI measures the level of blood flow to areas of the brain associated with mood and behaviour, and the participant will be asked to complete two behavioural games while they are in the scanner. During the scan, the participant will be required to lie on a table within the cylindrical tube of the MRI scanner in order to complete the scan. This will result in limited movement for the duration of the scan. The scan will take approximately 60 minutes.
Behavioral: Behavioural Games — The participant will be asked to complete two behavioural games inside the scanner. One of these games includes a monetary payout. They will be given instructions about these tasks outside of the scanner.

SUMMARY:
Major Depressive Disorder (MDD) is a very common illness that is usually treated with antidepressant medication. Depression can be caused by many things such as childhood experiences, genetics, and changes in the way the body and brain function. It is most likely caused by a combination of several of these factors. The prevalence of suicide attempt in Major Depressive Disorder (MDD) is about 20%. Risk for suicide attempt can be increased by many things such as negative life events, genetics, and changes in the way the body and brain function. It is most likely caused by a combination of several of these factors.

In this study, the investigators will be collecting detailed information about participants' psychiatric history and depression symptoms, as well as brain scans. The goal is to use this information to help us determine what predicts suicide attempt history.

ELIGIBILITY:
3.2 Inclusion Criteria

Depressed Participants:

1. Between the ages of 18 and 65 years old.
2. Capable of giving voluntary and informed consent.
3. Fluent in English.
4. Meet DSM-5 criteria for single or recurrent Major Depressive Disorder (current major depressive episode), confirmed via the Mini-International Neuropsychiatric Interview (MINI 6.086).
5. Moderate to severe depression severity, defined as a 17-item Hamilton Depression Rating Scale87 score ≥ 17.
6. Have had no initiation or dose change in any psychotropic medication in the four weeks prior to screening, as confirmed by the Antidepressant Treatment History Form (ATHF88).
7. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study.
8. Can adhere to the study schedule.
9. Either a history of or no lifetime history of suicide attempt, confirmed via the Mini-International Neuropsychiatric Interview (MINI 6.086).

Nondepressed Participants:

1. Between the ages of 18 and 65 years old.
2. Capable of giving voluntary and informed consent.
3. Fluent in English.
4. No current or lifetime history of psychiatric diagnoses or suicidality, confirmed via the MINI 6.086.
5. Absent/non-clinical depression severity, defined as a 17-item Hamilton Depression Rating Scale87 < 8.
6. No history of antidepressant use, as measured by the ATHF88.

3.3 Exclusion Criteria

All Participants:

1. Are pregnant/lactating.
2. A MINI-confirmed diagnosis of major depressive disorder in people with bipolar disorder.
3. Other major medical comorbidities requiring immediate investigation or treatment, cardiac pacemaker, or implanted medication pump.
4. Lifetime history of psychosis, confirmed by the MINI 6.086, including schizophrenia, schizoaffective disorder, delusional disorder, or current psychotic symptoms.
5. Drug abuse or dependence within the last 6 months, excluding caffeine and nicotine.
6. Presence of contraindications for MRI, including metallic implants.
7. Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, dementia, significant head trauma with loss of consciousness for greater than or equal to 5 minutes.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People will be assessed for a major depressive episode and history of suicide attempt. There will be three samples enrolled in this study:
  * Group 1: 50 healthy controls, or people who do not have depression.
  * Group 2: 50 people diagnosed with MDD and a history of suicide attempt
  * Group 3: 50 people diagnosed with MDD without a history of suicide attempt.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
fMRI Markers for Suicide Risk | Through study completion, an average of 1 week
  Potential fMRI brain activity for suicide risk using participants' brain scans

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Dunlop, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada